CLINICAL TRIAL: NCT00478998
Title: Phase II Study Comparing Two Groups of Patients Undergoing ESWL Treated With Ureteral Stents Versus Expulsion Therapy With Tamsulosin
Brief Title: Comparing Patients After ESWL Treated With Ureteral Stents Versus Expulsion Therapy With Tamsulosin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 890pal- HMO-CTIL
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2007-05-25 (Estimated); Status verified 2007-05

CONDITIONS: Upper Tract Ureterolithiasis
Keywords: expulsion therapy; tamsulosin; ureterolithiasis; stents
MeSH Terms: conditions — Ureterolithiasis | interventions — Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tamsulosin

SUMMARY:
The purpose of this study is to see whether patients undergoing ESWL, for upper tract urinary stones between 1.5-2.0cm, may be treated by expulsion therapy(Tamsulosin) instead of inserting ureteral stents .

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 yrs of age.
* Single urolithiasis up to 2 cm.
* Kidney/ureters that haven't undergone previous ESWL or stent insertion.
* Normal renal function (creatinine below 100mmo1/1).
* Sterile urine culture.
* Normal CBC, blood electrolytes and coagulation studies.
* Radioopaque stones.

Exclusion Criteria:

* More than one stone per kidney unit.
* Patients receiving steroids, NSAIDS, calcium channel blockers or alpha blockers on a regular basis.
* Anatomical anomalies or uromechanical obstruction.
* Single kidney.
* Cystinuria.
* Soldiers or pregnant women.
* Patients under 18 year

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
stone status at 3 month .
stone free

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Duvdevani, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel